CLINICAL TRIAL: NCT03759990
Title: A Comparison of Morbidly Obese and Lean
Brief Title: Tracheal Intubation in Morbidly Obese (BMI>35) and in Lean (BMI<30) Patients Using McGrath MAC X-Blade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KOU-KAEK 2018 - 202
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Obesity, Morbid
Keywords: videolaryngoscope; Airtraq; McGrath MAC; Morbid obesity; intubation
MeSH Terms: conditions — Obesity, Morbid | interventions — Adiposity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- insertion time (Active Comparator)
  Interventions: Device: lean; Device: obese
- intubation time (Active Comparator)
  Interventions: Device: lean; Device: obese

INTERVENTIONS:
Device: lean — Videolaryngoscope used in intubation
Device: obese — Videolaryngoscope used in intubation

SUMMARY:
80 lean (BMI<35) and morbidly obese (BMI>35) patients undergoing elective surgery were enrolled in this prospective ransomİzed study were intubated using McGrath MAC X-Blade. The demographic and airway variables of patients and insertion and intubation times with these dievices, need for optimisation maneuvers, hemodynamic changes and minör postoperative complications were recorded.

DETAILED DESCRIPTION:
80 lean (BMI<35) and morbidly obese (BMI>35) patients undergoing elective surgery were enrolled in this prospective ransomİzed study were intubated using McGrath MAC X-Blade. The demographic and airway variables of patients were recorded. Airway management variables Cormack-Lehan grades, insertion and intubation times, need for optimization maneuvers ( cricoid pressure, re-inserting, drawback) , hemodynamic changes in heart rate , blood pressure and minor postoperative complications such as sore throat, dysphasia, hoarseness were recorded.

ELIGIBILITY:
Inclusion Criteria: > 18 age <65 age

* bmı 35

  * undergoing elective surgery requiring endotracheal intubation

Exclusion Criteria: -pregnant

* <18 and >65 years of age
* bmı<35
* upper respiratory tract infection past ten days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
intubation time | 2 months

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University School of Medicine, Kocaeli
  - Kocaeli University Medical Faculty, Kocaeli

IPD SHARING:
Plan to Share IPD: No